CLINICAL TRIAL: NCT03029507
Title: An Acceptance and Commitment Therapy (ACT)-Enhanced Weight Management and Fitness Program for Navy Personnel
Brief Title: An ACT-enhanced Weight Management and Fitness Program for Navy Personnel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H160150
Record Dates: First submitted 2017-01-04; First posted 2017-01-24 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Military; Acceptance and Commitment Therapy; Overweight; Weight-management; Navy Personnel; Fitness
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT enhanced ShipShape (ACT +SS) (Experimental): The ACT+SS intervention will be delivered in 8 1.5-hour weekly group sessions. The ACT
  +SS protocol integrates ACT concepts and strategies within the existing standard SS protocol.
  Interventions: Behavioral: ACT Enhanced ShipShape
- Standard ShipShape (SS) (Active Comparator): Standard ShipShape (SS) The standard SS-only protocol will be delivered in 8 1.5-hour weekly group psychoeducation sessions.
  Interventions: Behavioral: Standard ShipShape (SS)

INTERVENTIONS:
Behavioral: ACT Enhanced ShipShape — The ACT components focus on: a) thoughts, feelings, and bodily sensations that are often present in the context of efforts to lose weight or improve fitness; b) limitations of previous efforts to control or eliminate negative thoughts or emotions, stress, or food cravings; c) changing expectations and goals from elimination of stress or cravings to living as well as possible with such feelings; d) mindfulness exercises to increase awareness of experiences; and e) identification of personal values and setting and pursuing values-consistent goals in order to achieve improved quality of life.
  Arms: ACT enhanced ShipShape (ACT +SS)
Behavioral: Standard ShipShape (SS) — The materials and format of the Standard SS-only protocol are based on recommendations from the Navy and Marine Corps Public Health Center. These include: a) education for nutrition and physical activity; b) creating and documenting goals for weight loss and physical fitness; c) a food diary to track eating habits throughout the program; d) developing behavioral strategies to initiate/maintain an exercise program; e) monitoring of physical activity (pedometer provided by the study); and f) identifying and overcoming personal triggers for over-eating.
  Arms: Standard ShipShape (SS)

SUMMARY:
The proposed study is a cohort-randomized controlled trial of Acceptance and Commitment Therapy-enhanced ShipShape (ACT+SS) compared to the standard ShipShape-only program, for overweight or obese Navy personnel. As a result of COVID-19, this study is now being conducted virtually.

DETAILED DESCRIPTION:
The proposed study is a cohort-randomized controlled trial of ACT-enhanced SS (ACT+SS) compared to the SS-only program. Cohorts of Navy personnel who are failing or at risk of failing the body composition assessment (BCA) or who are overweight/obese will be randomized to receive 8 weekly ACT+SS intervention groups or 8 weekly SS-only intervention groups. The scientific aims are to: 1) determine the effectiveness of ACT+SS compared to the SS-only program; 2) examine psychological flexibility as a mechanism underlying intervention response; and 3) explore potential moderators of intervention response. The primary outcome is weight loss.

Secondary outcomes include BMI, body fat %, indices of physical activity, problem eating, functioning and quality of life, emotional functioning and indices of psychological flexibility, measured at baseline, mid- and post-intervention, and 3- and 6-month follow-up and self- reported BCA status at 6-month follow-up. The investigators have purposefully designed a cohort-randomized trial with interventions that are pragmatically implemented in a real-life military setting, and outcomes that are immediately relevant to service members and leadership. The cohort randomization is essential to the feasibility and acceptability of the research in this setting. The military-relevant and generalizable findings are more likely to have impact within the military. SS provides an ideal comparison arm that is the current standard of practice in the Navy. Integrating ACT with SS in this setting overcomes many of the logistical, practical, chain-of-command, and other challenges that have typically impeded research in the military. The investigators have thoughtfully selected primary and secondary outcomes that are theoretically linked, and additional assessments that are empirically-based and will allow better understanding of mediators and moderators of intervention response in Navy personnel. Due to Covid-19 we have adapted the interventions to be administered virtually.

ELIGIBILITY:
Inclusion Criteria:

* Navy Personnel who are overweight/obese or have failed or are at risk of failing the BCA
* 18-69 years of age
* Willingness to participate in the study

Exclusion Criteria:

* Any physical limitations (injuries, pregnancy, etc.) that preclude engagement in the physical fitness activities

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in weight from baseline | Outcome measures will be completed at study baseline (week 1), mid treatment ( week 4), post-treatment (week 8), and 3 and 6 month follow-up post-treatment.

SECONDARY OUTCOMES:
Change in Three-Factor Eating Questionnaire (TFEQ-R18) score | Outcome measures will be completed at study baseline (week 1), mid treatment ( week 4), post-treatment (week 8), and 3 and 6 month follow-up post-treatment.
Change in weight related Acceptance and Action Questionnaire for Weight-Related Difficulties-Revised (AAQW-R) | Outcome measures will be completed at study baseline (week 1), mid treatment ( week 4), post-treatment (week 8), and 3 and 6 month follow-up post-treatment.
Change in Satisfaction with Life Scale (SWLS) | Outcome measures will be completed at study baseline (week 1), mid treatment ( week 4), post-treatment (week 8), and 3 and 6 month follow-up post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Niloofar Afari, PhD, Principal Investigator — Veterans Medical Research Foundation
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Veterans Medical Research Foundation, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Dochat C, Afari N, Wooldridge JS, Herbert MS, Gasperi M, Lillis J. Confirmatory Factor Analysis of the Acceptance and Action Questionnaire for Weight-Related Difficulties-Revised (AAQW-R) in a United States Sample of Adults with Overweight and Obesity. J Contextual Behav Sci. 2020 Jan;15:189-196. doi: 10.1016/j.jcbs.2020.01.006. Epub 2020 Jan 10. PMID 32257780
- [Background] Afari N, Cuneo JG, Herbert M, Miller I, Webb-Murphy J, Delaney E, Peters J, Materna K, Miggantz E, Godino J, Golshan S, Wisbach G. Design for a cohort-randomized trial of an acceptance and commitment therapy-enhanced weight management and fitness program for Navy personnel. Contemp Clin Trials Commun. 2019 Jul 10;15:100408. doi: 10.1016/j.conctc.2019.100408. eCollection 2019 Sep. PMID 31338482
- [Derived] Afari N, Yarish NM, Wooldridge JS, Materna K, Hernandez J, Blanco BH, Camodeca AL, Peters JJ, Herbert MS. Lessons Learned From Transition of an In-Person to a Virtual Randomized Controlled Trial for Weight and Fitness Concerns in Active-Duty Service Members: Survey Study. J Med Internet Res. 2022 Nov 10;24(11):e37797. doi: 10.2196/37797. PMID 36201851